CLINICAL TRIAL: NCT01595581
Title: The Effects of Acute Testosterone Administration in Men on Muscle Mass, Strength, and Physical Function Following ACL Reconstructive Surgery
Brief Title: Testosterone Administration and ACL Reconstruction in Men
Acronym: TACL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Boston University (Other); University of Oregon (Other)
Responsible Party: Principal Investigator, Todd Schroeder, Assistant Professor of Clinical Physical Therapy, University of Southern California
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-11-00649
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Muscle Atrophy; ACL Reconstruction; Trauma; Osteoarthritis
Keywords: Testosterone; ACL Reconstruction; Clinical outcomes; Lean mass; Strength; Muscle atrophy
MeSH Terms: conditions — Muscular Atrophy; Wounds and Injuries; Osteoarthritis | interventions — Testosterone; testosterone enanthate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Testosterone (Experimental): Weekly injection of testosterone enanthate 200mg
  Interventions: Drug: Testosterone
- Placebo (Placebo Comparator): Weekly injection of saline as the placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone — 8 weeks of testosterone administration beginning 2 weeks before ACL surgery
  Other Names: testosterone enanthate
  Arms: Testosterone
Drug: Placebo — 8 weeks of saline administration beginning 2 weeks before ACL surgery
  Other Names: saline
  Arms: Placebo

SUMMARY:
This study is being done to test whether taking testosterone can prevent loss of muscle mass and strength due to anterior cruciate ligament (ACL) reconstructive surgery. Testosterone is the principal male sex hormone and an anabolic (muscle promoting) steroid. It is essential for the development of male reproductive tissues and promotes increased muscle, bone mass, and the growth of body hair.

The investigators hope to learn whether testosterone given before and after ACL reconstructive surgery will increase muscle mass and strength and potentially improve recovery time following surgery.

DETAILED DESCRIPTION:
Overall Objective: The overall objective of this study is to determine if 8 weeks of testosterone first administered 2 weeks prior to surgery, can improve the outcome of anterior cruciate ligament (ACL) reconstruction.

Overall Hypothesis: Standard-of-care rehabilitation with the addition of testosterone administration will augment muscle mass, strength, and physical function following ACL reconstructive surgery compared to standard rehabilitation alone.

Significance: Muscle mass and strength are greatly reduced following ACL surgery. The investigators hypothesize that administration of testosterone will minimize these reductions or potentially increase muscle mass and strength. In doing so, testosterone may hasten a patient's return to physical activity. If testosterone improves recovery after ACL surgery, the same treatment may be used for other injuries that involve trauma and muscle atrophy. Furthermore, this study will examine the effect of trauma with or without testosterone on myogenic regulators in muscle tissue taken during ACL surgery-providing possible mechanistic insights for the clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* A complete ACL tear as visualized on MRI
* The ACL injury can be either "isolated" or combined with one or several of the following injuries visualized on MRI and/or arthroscopy:
* a meniscus tear that is either left untreated or treated with a partial resection
* a small, stable meniscus tear treated with fixation, but with the fixation not interfering with the rehabilitation protocol
* cartilage changes verified on MRI with an arthroscopically determined intact surface.
* A radiographic examination with normal joint status or combined with either one of the following findings:
* a small-avulsed fragment located laterally, usually described as a Segond fracture, JSN grade 1 or osteophytes grade 1 as determined by the OARSI atlas15

Exclusion Criteria:

* Previous major knee injury or knee surgery
* Associated posterior cruciate ligament (PCL) or medical collateral ligament (MCL) injury grade III
* Concomitant severe injury to contra-lateral knee
* Injury to the lateral/posterolateral ligament complex with significantly increased laxity
* Unstable longitudinal meniscus tear that requires repair and where the following postoperative treatment (we.e. bracing and limited range of motion) interferes with the rehabilitation protocol
* Bi-compartmental extensive meniscus resections
* Cartilage injury representing a full thickness loss down to bone
* Total rupture of MCL/LCL as visualized on MRI.
* History of deep vein thrombosis (DVT) or a disorder of the coagulative system
* Claustrophobia
* Prior or current use of anabolic steroids
* General systemic disease affecting physical function
* Chromosomal disorders
* Medications that interfere with testosterone production or function, including but not limited to 5α-reductase inhibitors
* Any other condition or treatment interfering with the completion of the trial

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Schroeder, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu B, Lorezanza D, Badash I, Berger M, Lane C, Sum JC, Hatch GF 3rd, Schroeder ET. Perioperative Testosterone Supplementation Increases Lean Mass in Healthy Men Undergoing Anterior Cruciate Ligament Reconstruction: A Randomized Controlled Trial. Orthop J Sports Med. 2017 Aug 9;5(8):2325967117722794. doi: 10.1177/2325967117722794. eCollection 2017 Aug. PMID 28840147
- [Derived] Wu BW, Berger M, Sum JC, Hatch GF 3rd, Schroeder ET. Randomized control trial to evaluate the effects of acute testosterone administration in men on muscle mass, strength, and physical function following ACL reconstructive surgery: rationale, design, methods. BMC Surg. 2014 Dec 6;14:102. doi: 10.1186/1471-2482-14-102. PMID 25481088

RESULTS

PARTICIPANT FLOW:
Groups:
- Testosterone: Testosterone: 8 weeks supraphysiologic dose testosterone enanthate
- Placebo: Saline: Placebo for 8 weeks
Period: Overall Study
Arm/Group | Testosterone | Placebo
Started | 7 | 7
Completed | 6 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Testosterone: Testosterone: 8 weeks 200mg dose testosterone enanthate
- Total: Total of all reporting groups
Arm/Group | Testosterone | Placebo | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (9.3) | 26.2 (4.1) | 28.2 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 7 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Recruited from the Los Angeles area
  participants
    United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Changes in Lean Mass
Description: Relative changes in lean mass from 2 weeks prior to surgery to 6 weeks, 12 weeks, and 24 weeks following surgery between the two groups.
Time Frame: 6, 12, and 24 weeks post operative
Population: Region of enrollment from the Los Angeles area.
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Testosterone: Testosterone: 8 weeks supraphysiologic dose testosterone enanthate. Ethnicity: 4 White, 2 Asian, 1 Black
- Placebo: Saline: Placebo for 8 weeks
  Ethnicity: 4 White, 1 Asian, 2 Hispanic
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 6 | 7
kg
  6 weeks post op | 2.8 (1.7) | -0.1 (1.5)
  12 weeks post op | 2.16 (3.48) | 0.01 (1.08)
  24 weeks post op | 2.13 (5.3) | 1.05 (1.18)
Statistical Analysis 1: Comparison: Testosterone vs Placebo; Power was estimated for change in lean mass of 3.0 plus or minus 1.5 kg in healthy men receiving testosterone. Using a significance level of 0.05 and a power of 0.80, a sample size of 6 participants per group was calculated. This statistical analysis applies to lean mass in participants 6 weeks post operative; Test type: Other — Mann-Whitney U test for continuous variables and Fisher exact test for categorical variables; p = 0.35, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 2.9, Standard Deviation 1.5
Statistical Analysis 2: Comparison: Testosterone vs Placebo; Power was estimated for change in lean mass of 3.0 plus or minus 1.5 kg in healthy men receiving testosterone. Using a significance level of 0.05 and a power of 0.80, a sample size of 6 participants per group was calculated. This statistical analysis applies to lean mass in participants 12 weeks post operative; Test type: Other; p = 0.48, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 2.17, Standard Deviation 2
Statistical Analysis 3: Comparison: Testosterone vs Placebo; Power was estimated for change in lean mass of 3.0 plus or minus 1.5 kg in healthy men receiving testosterone. Using a significance level of 0.05 and a power of 0.80, a sample size of 6 participants per group was calculated. This statistical analysis applies to lean mass in participants 24 weeks post operative; Test type: Other; p = 0.74, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 1.08, Standard Deviation 15

2. Secondary Outcome: KOOS Scores
Description: Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) from 2 weeks prior to surgery to 6, 12, and 24 weeks post surgery.
  KOOS is scored from 0 to 100 with 0 representing extreme knee problems and 100 representing normal knee function.
Time Frame: 6 weeks, 12 weeks, 24 weeks post surgery
Population: Region of enrollment from the Los Angeles area.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 6 | 7
score on a scale
  6 weeks post op | 63.2 (10.6) | 65.5 (13)
  12 weeks post op | 76.7 (9.9) | 73.2 (15)
  24 weeks post op | 84 (9.4) | 86.6 (8.3)

3. Secondary Outcome: Strength
Description: Changes in muscle strength from the start of rehabilitation to 6, 12, and 24 weeks following surgery between the two groups in the injured limb.
Time Frame: 6, 12, and 24 weeks post surgery
Population: Region of enrollment from the Los Angeles area.
Measure: Mean (Standard Deviation); unit: Nm
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 6 | 7
Nm
  6 weeks post op | -53.5 (35.8) | -33.4 (37.4)
  12 weeks post op | -18.3 (52.7) | -6.6 (40.3)
  24 weeks post op | 19.2 (60.9) | 19.0 (33.9)

ADVERSE EVENTS:
Time Frame: Trough the study completion (24-weeks).
Description: All subjects were monitored/assessed for adverse events.
Arm/Group | Testosterone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes